CLINICAL TRIAL: NCT00562588
Title: EARLY: Prospective, Randomised, National, Multi-centre, Open-label, Blinded Endpoint Study to Compare Aggrenox b.i.d. (200 mg Dipyridamole MR + 25 mg Acetylsalicylic Acid) When Started Within 24 Hours of Stroke Onset on an Acute Stroke Unit, and Aggrenox b.i.d. When Started After a 7-day Therapy With ASA 100 mg Once Daily Outside Off an Acute Stroke Unit, in Symptomatic Ischaemic Stroke Patients Over a Three Months Treatment Period an Exploratory Study
Brief Title: EARLY 3-months Aggrenox Treatment Started Within 24 Hrs of Ischemic Stroke Onset vs. After One Week 100 mg ASA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 9.182
Record Dates: First submitted 2007-07-06; First posted 2007-11-22 (Estimated); Results first posted 2010-03-11 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-01

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Drug: Aggrenox bid (ASA 25mg/Dipyridamole ER 200mg)
Drug: ASA 100 mg qd

SUMMARY:
German stroke units are hesitating to use Aggrenox for secondary ischaemic stroke / transient ischaemic attack (TIA) prevention in a sub-acute treatment setting. They argue that clinical experience with sub-acute Aggrenox treatment is limited and poorly documented when compared with sub-acute acetylsalicylic acid (ASA) treatment. However, long term treatment (started after 3-6 months after stroke/TIA) with Aggrenox was safe and superior to ASA treatment in preventing recurrent strokes. There is no evidence for ASA to prevent from neurological progression after stroke during the first 3 months. Results from a cohort study suggest that starting Aggrenox within 72 hours after stroke predicts clinical improvement in the National Institute of Health Stroke Scale (NIHSS) at discharge from the hospital. Dipyridamole suppresses acute inflammatory responses to stroke.

This study is designed to investigate the tolerability and efficacy of a secondary stroke prevention treatment with Aggrenox when initiated within 24 hours of stroke onset on a stroke unit compared to later initiation after a 7 day ASA treatment and outside off a stroke unit setting.

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of ischaemic stroke causing a measurable neurological deficit defined as impairment of language, motor function, cognition and/or gaze, vision or neglect. Symptoms must be distinguishable from an episode of generalised ischaemia (i.e. syncope), seizure, or migraine disorder.

Main inclusion criteria:

* Patients at risk of stroke who have had transient ischaemia of the brain or completed ischaemic stroke due to thrombosis
* Symptoms of ischaemic attack began less than 24 hours prior to study medication start, are to be present for at least 30 minutes and have not significantly improved before start of treatment
* Patients are eligible for platelet inhibiting treatment
* National Institute of Health Stroke Scale (NIHSS) between 5 and 20 (at pre-screening and screening)
* Actual Modified Rankin Scale (mRS) (at baseline) is worse than retrospective mRS (before stroke)
* A contraindication for stroke lysis is given
* Patients are able to give (at least oral) informed consent and to swallow either medication

Exclusion Criteria:

* Hypersensitivity to any of the components of the product or salicylates.
* Patients with active gastric or duodenal ulcers or with bleeding disorders.
* Pregnancy during the third trimester.
* Lysis therapy.
* A platelet inhibiting therapy with Acetylsalicylic Acid (ASA) doses of more than 100 mg per day, or with clopidogrel of any dose has been planned or started.
* Time of onset of stroke symptoms is unknown (when a stroke happened during night-/sleeping time, bedtime is assumed as time of onset)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 9.182.1 Boehringer Ingelheim Investigational Site, Bad Homburg, Germany

REFERENCES:
- [Derived] Dengler R, Diener HC, Schwartz A, Grond M, Schumacher H, Machnig T, Eschenfelder CC, Leonard J, Weissenborn K, Kastrup A, Haberl R; EARLY Investigators. Early treatment with aspirin plus extended-release dipyridamole for transient ischaemic attack or ischaemic stroke within 24 h of symptom onset (EARLY trial): a randomised, open-label, blinded-endpoint trial. Lancet Neurol. 2010 Feb;9(2):159-66. doi: 10.1016/S1474-4422(09)70361-8. Epub 2010 Jan 7. PMID 20060783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 551 patients enrolled, 548 randomized, 543 treated; analysis is based on treated patients
Groups:
- Aspirin for 7 Days, Followed by Aggrenox: ASA 100 mg qd for 7 days, followed by Aggrenox (dipyridamole 200mg + ASA 25mg) b.i.d
- Aggrenox: Aggrenox (dipyridamole 200mg + ASA 25mg) b.i.d
Period: Overall Study
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Started | 260 | 283
Completed | 168 | 184
Not Completed | 92 | 99
Not completed — Adverse Event | 40 | 58
Not completed — Protocol Violation | 30 | 26
Not completed — Lost to Follow-up | 12 | 4
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox | Total
Number analyzed (Participants) | 260 | 283 | 543
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.3 (11.5) | 66.5 (11.4) | 67.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 109 | 204
  Male | 165 | 174 | 339

OUTCOME MEASURES:

1. Primary Outcome: Telephone Modified Rankin Scale (Centralised, Blinded Assessment)
Description: The modified Rankin Scale (mRS) is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0-6, running from perfect health without symptoms to death. Best value - 0 (No symptoms), worst value - 6 (Dead)
Time Frame: 90 days
Population: FAS which included all randomised patients who had follow up data available (mRS or NIHSS) or who were dead.
Measure: Number; unit: participants
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 254 | 273
participants
  0 | 58 | 70
  1 | 75 | 84
  2 | 50 | 62
  3 | 30 | 16
  4 | 31 | 32
  5 | 6 | 4
  6 | 4 | 5
Statistical Analysis 1: Comparison: Aspirin for 7 Days, Followed by Aggrenox vs Aggrenox; The primary endpoint tele-mRS on day 90 was available in 527 of 543 treated patients (97.1%); Test type: Superiority or Other; p = 0.683, Regression, Logistic; Odds Ratio (OR) = 1.067, 95% CI [0.78 to 1.461]

2. Secondary Outcome: Change From Baseline in NIHSS (National Institutes of Health Stroke Scale)
Description: The NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from 0 (no deficit) to 42 (dead)
Time Frame: Baseline and 90 days
Population: FAS which included all randomised patients who had follow up data available (mRS or NIHSS) or who were dead.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 238 | 262
Units on a scale | -2 [-4 to 0] | -2 [-3 to 0]
Statistical Analysis 1: Comparison: Aspirin for 7 Days, Followed by Aggrenox vs Aggrenox; Early treatment initiation (immediately after the index event) with Aggrenox was compared to late initiation of Aggrenox after 7 days of treatment with ASA mono; Test type: Superiority or Other; p = 0.607, ANCOVA; ANCOVA with factors for treatment, age, weight, baseline SBP, diabetes, previous stroke and baseline NIHSS

3. Secondary Outcome: Patients With Relevant Event (Death, Non-fatal Stroke, Transient Ischaemic Attack (TIA), Myocardial Infarction (MI), Bleeding)
Time Frame: 90 days
Population: FAS which included all randomised patients who had follow up data available (mRS or NIHSS) or who were dead.
Measure: Number; unit: participants
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 260 | 283
participants | 38 | 28
Statistical Analysis 1: Comparison: Aspirin for 7 Days, Followed by Aggrenox vs Aggrenox; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.202, Cox proportional hazards model; Hazard Ratio (HR) = 0.725, 95% CI [0.442 to 1.189]

4. Secondary Outcome: Telephone Modified Rankin Scale (Centralised, Blinded Assessment) at Day 8
Description: as for outcome 1
Time Frame: 8 days
Population: FAS which included all randomised patients who had follow up data available (mRS or NIHSS) or who were dead.
Measure: Number; unit: participants
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 254 | 273
participants
  0 | 46 | 47
  1 | 59 | 74
  2 | 42 | 52
  3 | 39 | 38
  4 | 51 | 44
  5 | 12 | 8
  6 | 0 | 2
  Missing | 5 | 8

5. Secondary Outcome: Change From Baseline in NIHSS (National Institutes of Health Stroke Scale) at Day 8
Description: as for outcome 2
Time Frame: Baseline and 8 days
Population: FAS which included all randomised patients who had follow up data available (mRS or NIHSS) or who were dead.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 236 | 255
units on a scale | -1.0 [-3.0 to 0.0] | -1.0 [-3.0 to 0.0]

6. Secondary Outcome: Change of Special Biochemical Laboratory Value- CRP
Description: Changes of special biochemical laboratory values (CRP) from baseline to day 8 - centralised, blinded assessment by a specialised central clinical laboratory
Time Frame: 8 days
Population: FAS which included all randomised patients who had follow up data available (mRS or NIHSS) or who were dead.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 213 | 212
mg/L | 1.27 [1.06 to 1.52] | 1.17 [1.00 to 1.38]

7. Secondary Outcome: Change of Special Biochemical Laboratory Value- MMP-9
Description: Changes of special biochemical laboratory value (MMP-9) from baseline to day 8 - centralised, blinded assessment by a specialised central clinical laboratory
Time Frame: 8 days
Population: FAS which included all randomised patients who had follow up data available (mRS or NIHSS) or who were dead.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 213 | 212
ng/mL | 0.974 [0.884 to 1.07] | 0.983 [0.89 to 1.08]

8. Secondary Outcome: Change of Special Biochemical Laboratory Value - MCP-1
Description: Changes of special biochemical laboratory value (MCP-1) from baseline to day 8 - centralised, blinded assessment by a specialised central clinical laboratory
Time Frame: 8 days
Population: FAS which included all randomised patients who had follow up data available (mRS or NIHSS) or who were dead.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 213 | 212
µg/mL | 1.06 [1.01 to 1.10] | 1.08 [1.03 to 1.13]

9. Secondary Outcome: Change From Baseline in FLAIR (Fluid-Attenuated Inversion Recovery) at Day 8
Description: MRI was performed to assess growth in stroke lesion volume by fluid-attenuated inversion recovery (FLAIR).
Time Frame: Baseline and day 8
Population: Full Analysis Set - included all randomised patients who had value in FLAIR at baseline and day 8.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 116 | 111
mL | 0.4100 [0.1050 to 2.0450] | 0.3300 [0.0200 to 1.3500]

10. Secondary Outcome: Change From Baseline in FLAIR (Fluid-Attenuated Inversion Recovery) at Day 90.
Description: MRI was performed to assess growth in stroke lesion volume by fluid-attenuated inversion recovery (FLAIR).
Time Frame: Baseline and day 90
Population: Full Analysis Set - included all randomised patients who had value in FLAIR at baseline and day 90.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 101 | 90
mL | 0.1900 [0.0000 to 1.1400] | 0.1150 [0.0000 to 0.9000]

11. Secondary Outcome: Change From Baseline in DWI (Diffuse-Weighted Imaging) at Day 8
Description: MRI was performed to assess growth in stroke lesion volume by diffusion-weighted imaging (DWI). DWI was to give evidence of the development of the ischaemic lesion corresponding to the evolved stroke.
Time Frame: Baseline and day 8
Population: Full Analysis Set - included all randomised patients who had value in DWI at baseline and day 8.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 120 | 117
mL | -0.0600 [-0.7050 to 0.5650] | 0.0000 [-0.5000 to 0.3000]

12. Secondary Outcome: Change From Baseline in DWI (Diffuse-Weighted Imaging) at Day 90
Description: as for outcome 11
Time Frame: Baseline and day 90
Population: Full Analysis Set - included all randomised patients who had value in DWI at baseline and day 90.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Number analyzed (Participants) | 80 | 70
mL | -0.8400 [-2.0850 to -0.3550] | -0.7100 [-1.9300 to -0.2600]

ADVERSE EVENTS:
Time Frame: Up to 90 days
Description: From first drug intake until date of last drug intake
Arm/Group | Aspirin for 7 Days, Followed by Aggrenox | Aggrenox
Serious Adverse Events (participants affected / at risk) | 48/260 | 45/283
Other Adverse Events (participants affected / at risk) | 60/260 | 119/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin for 7 Days, Followed by Aggrenox (N=260) | Aggrenox (N=283)
Cerebrovascular accident (Nervous system disorders) | 15 | 5
Carotid artery stenosis (Nervous system disorders) | 5 | 2
Transient ischaemic attack (Nervous system disorders) | 4 | 2
Ischaemic stroke (Nervous system disorders) | 3 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Hemiplegia (Nervous system disorders) | 1 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 2
Status epilepticus (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Basilar artery thrombosis (Nervous system disorders) | 1 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Diabetic coma (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hyponatraemic encephalopathy (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 3
Myocardial infarction (Cardiac disorders) | 1 | 4
Cardiac failure (Cardiac disorders) | 1 | 3
Aortic valve stenosis (Cardiac disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular dyskinesia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Appendicitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 3 | 3
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Arterial repair (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin for 7 Days, Followed by Aggrenox (N=260) | Aggrenox (N=283)
Headache (Nervous system disorders) | 53 | 105
Nausea (Gastrointestinal disorders) | 14 | 29
Vomiting (Gastrointestinal disorders) | 10 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.